CLINICAL TRIAL: NCT06754826
Title: Effectiveness of AI-Generated Questions and Feedback in Learning Diagnostic Reasoning: An Experimental Study
Brief Title: Learning Diagnostic Reasoning Through AI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Yavuz Selim KIYAK, Principal Investigator, Gazi University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2024 - 2019
Record Dates: First submitted 2024-12-19; First posted 2025-01-01 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Artificial Intelligence (AI); Clinical Reasoning; Medical Education; Feedback
Keywords: artificial intelligence; diagnostic reasoning; clinical reasoning; medical education; feedback

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): The group who receives AI-generated questions and feedback related to five abdominal pain diagnoses.
  Interventions: Other: AI-generated questions and feedback as a spaced repetition
- Control Group (No Intervention): The group who does not receive AI-generated questions and feedback related to five abdominal pain diagnoses.

INTERVENTIONS:
Other: AI-generated questions and feedback as a spaced repetition — Participants in the intervention group will undergo structured learning sessions consisted of AI-generated questions and feedback as a spaced repetition.
  Arms: Intervention Group

SUMMARY:
This experiment aims to determine the effect of AI-generated questions and feedback on diagnostic reasoning in preclinical medical students.

Main Research Question:

What is the effect of AI-generated questions and feedback on diagnostic reasoning skills in preclinical medical students?

DETAILED DESCRIPTION:
This study involves a two groups:

1. Intervention Group: Medical students will receive AI-generated questions and feedback related to five abdominal pain diagnoses.
2. Control Group: Medical students will not receive any intervention. Participants in the intervention group will undergo structured learning sessions consisted of AI-generated questions and feedback as a spaced repetition. Control group will not attend these sessions; they only receive their usual medical training.

The diagnostic reasoning performance will be assessed using a video-based Objective Structured Clinical Examination: OSVE (Objective Structured Video Examination) where videos of "patient-doctor encounters are shown to students and questions related to the video clip are asked. Written answers are marked in a standardised manner."

ELIGIBILITY:
Inclusion Criteria:

Medical students in Gazi University Faculty of Medicine

Exclusion Criteria:

Medical students outside Gazi University Faculty of Medicine

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2025-01-27 (Actual); Primary Completion 2025-02-16 (Actual); Study Completion 2025-02-16 (Actual)

PRIMARY OUTCOMES:
Diagnostic Reasoning Performance | up to 30 days
  The diagnostic reasoning performance will be assessed using a video-based Objective Structured Clinical Examination: OSVE (Objective Structured Video Examination) where videos of "patient-doctor encounters are shown to students and questions related to the video clip are asked. Written answers are marked in a standardised manner."

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University Faculty of Medicine, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The dataset (containing information about correct and incorrect answers) will be shared without including participants' identifiable information (e.g., names). Identifiable data will be replaced with codes (e.g., Participant 1, Participant 2, etc.).
Access Criteria: The dataset will be publicly available.